CLINICAL TRIAL: NCT02259790
Title: Relative Bioavailability of Telmisartan 40 mg/Amlodipine 5 mg Fixed-dose Combination Tablet Compared to Concomitant Use of Its Mono-components (i.e., Telmisartan 40 mg Tablet and Amlodipine 5 mg Tablet in Concomitant Use) Following Oral Administration in Healthy Male Volunteers (an Open-label, Randomised, Single Dose, Two-way Crossover Study)
Brief Title: Bioavailability of Telmisartan/Amlodipine Fixed-dose Combination Compared to Its Mono-components in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1235.17
Record Dates: First submitted 2014-10-06; First posted 2014-10-09 (Estimated); Last update posted 2014-10-09 (Estimated); Status verified 2014-10

CONDITIONS: Healthy
MeSH Terms: interventions — Telmisartan; Amlodipine

ARMS (2):
- Telmisartan/amlodipine fixed-dose combination (Experimental)
  Interventions: Drug: Telmisartan/amlodipine fixed-dose combination tablet
- Telmisartan tablet and amlodipine tablet (Active Comparator)
  Interventions: Drug: Telmisartan; Drug: Amlodipine

INTERVENTIONS:
Drug: Telmisartan/amlodipine fixed-dose combination tablet
  Arms: Telmisartan/amlodipine fixed-dose combination
Drug: Telmisartan
  Arms: Telmisartan tablet and amlodipine tablet
Drug: Amlodipine
  Arms: Telmisartan tablet and amlodipine tablet

SUMMARY:
Study to investigate the relative bioavailability of fixed-dose combination tablet vs.

mono-components of telmisartan and amlodipine

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males according to the following criteria:

   Based upon a complete medical history, including the physical examination, vital signs (blood pressure, pulse rate and body temperature), 12-lead ECG, clinical laboratory tests, no finding of clinical relevance, no evidence of a clinically relevant concomitant disease
2. Age ≥20 and Age ≤35 years
3. Body weight ≥50 kg
4. BMI ≥17.6 and BMI ≤26.4 kg/m2 (Body Mass Index)
5. Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice

Exclusion Criteria:

1. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
2. Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
3. Chronic or relevant acute infections
4. Any clinical relevant findings of the laboratory test deviating from normal
5. Positive result for hepatitis B antigen, anti hepatitis C virus anti bodies, syphilitic test or HIV test
6. Surgery of gastrointestinal tract (except appendectomy)
7. History of relevant orthostatic hypotension (mean standing systolic blood pressure (SBP) varies by ≥20 mmHg from mean supine SBP or mean standing diastolic blood pressure (DBP) varies by ≥10 mmHg from mean supine DBP), fainting spells or blackouts
8. History of hepatic dysfunction (e.g. biliary cirrhosis, cholestasis)
9. History of serious renal dysfunction
10. History of bilateral renal artery stenosis or renal artery stenosis in a solitary kidney
11. History of cerebrovascular disorder
12. History of hyperkalemia
13. Known hypersensitivity to any component of the formulation, or to any other angiotensin II receptor antagonists, angiotensin converting enzyme or dihydropyridine
14. Intake of drugs with a long half-life (≥24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
15. Use of drugs which might reasonably influence the results of the trial based on the knowledge at the time of protocol preparation within 7 days prior to administration or during the trial
16. Participation in another trial with an investigational drug within 4 months or 6 half-lives of the investigational drug prior to administration
17. Smoker (≥20 cigarettes/day)
18. Alcohol abuse (60 g or more ethanol/day: ex. 3 middle-sized bottles of beer, 3 gous (equivalent to 540 mL) of sake)
19. Drug abuse
20. Blood donation (more than 100 mL within 4 weeks prior to administration or during the trial)
21. Excessive physical activities (within 1 week prior to administration or during the trial)
22. Intake of alcohol within 2 days prior to administration
23. Inability to comply with dietary regimen of study centre
24. Intake of any drugs/supplements with ingredient of hypericum perforatum or citrus fruits (e.g. grapefruits, Sevilla orange) within 5 days prior to administration
25. Inability to refrain from smoking on trial days
26. Any other volunteers whom, the principal investigator or sub investigator would not allow to participate in this study

Ages: 20 Years to 35 Years | Sex: Male
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2007-07; Primary Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz) | up to 144 hours after administration of study drug
Maximum measured concentration of the analyte in plasma (Cmax) | up to 144 hours after administration of study drug

SECONDARY OUTCOMES:
Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) | up to 144 hours after administration of study drug
Time from administration to the maximum concentration of the analyte in plasma (tmax) | up to 144 hours after administration of study drug
Terminal rate constant of the analyte in plasma (λz) | up to 144 hours after administration of study drug
Terminal half-life of the analyte in plasma (t1/2) | up to 144 hours after administration of study drug
Mean residence time of the analyte in the body after po administration (MRTpo) | up to 144 hours after administration of study drug
Number of subjects with adverse events | up to 56 days
Number of subjects with clinically significant changes in vital signs | up to 144 hours after administration of study drug
Number of subjects with clinically significant changes in 12-lead ECG (electrocardiogram) | up to 144 hours after administration of study drug
Number of subjects with clinically significant changes in laboratory tests | up to 144 hours after administration of study drug